CLINICAL TRIAL: NCT01877031
Title: Needle Guidance With Virtual Reality Augmented Ultrasound Versus Ultrasound Guidance Alone For Central Line Insertion: A Randomized Trial.
Brief Title: Virtual Reality With Ultrasound Versus Ultrasound For Central Line Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: University of Western Ontario, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: R-11-607
Record Dates: First submitted 2013-06-09; First posted 2013-06-13 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Central Line Complication
Keywords: central line; ultrasound guided central line insertion; virtual reality; augmented reality
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound (Active Comparator): Ultrasound only guidance of central line insertion - current standard of care.
  Interventions: Device: Ultrasound
- Virtual Reality (Experimental): Use of ultrasound plus virtual reality guidance to insert central line
  Interventions: Device: Virtual Reality

INTERVENTIONS:
Device: Virtual Reality — A magnetically tracked needle with an associated virtual image will be superimposed on the ultrasound image to give the user a better idea of the position of the needle.
  Other Names: Augmented reality
  Arms: Virtual Reality
Device: Ultrasound — Standard of Care - Ultrasound guided intervention
  Arms: Ultrasound

SUMMARY:
We aim to compare the use of ultrasound guidance alone versus a magnetically tracked needle to look at the time taken to place a central line, or specifically the time taken to place a needle in the internal jugular vein prior to utilizing the Seldinger technique to insert a central line.

DETAILED DESCRIPTION:
The purpose of this study is to examine the incremental benefit of a innovative, robust, intuitive and portable, virtual reality(VR) imaging platform capable of displaying a tracked virtual needle tip with path trajectory along with the real time ultrasound(US) image of an internal jugular vein compared to US imaging of the internal jugular vein alone to reduce the complications associated with insertion of central lines.

The studies primary outcome is the difference in time to insert a central line, from needle insertion to placement and confirmation of the wire in the internal jugular vein, compared to standard insertions using ultrasound guidance alone. Secondary outcomes will include the number of needle withdrawals, the incidence of carotid puncture and the incidence of pneumothorax. Finally, a subjective VAS rating of 1 to 10 for ease of insertion will be collected from participating anesthesiologists.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* Require a central line inserted in the left jugular vein
* Undergoing surgery

Exclusion Criteria:

* Contraindication to left jugular vein insertion (absent vein, infection at site)
* Permanent or temporary pacemaker
* Emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Time taken to insert needle | within 15 minutes
  Measure the time taken from needle on skin to blood in syringe

SECONDARY OUTCOMES:
Attempts | 15 minutes
  Measure the number of attempts taken to locate the internal jugular vein. Measured by the number of times the needle is advanced.
Carotid Puncture | within 24 hours
  Record if the carotid artery was hit (clinical)
Pneumothorax | 24 hours
  Monitor for pneumothorax after the procedure (clinical, Chest X-ray)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Bainbridge, MD FRCPC, Principal Investigator — Western University, Canada
Locations (1):
- London Health Sciences Center, London, Ontario, Canada